CLINICAL TRIAL: NCT00980187
Title: A Comparison of Indapamide SR 1.5 mg With Hydrochlorothiazide 25 mg, in Combination With an ACE-inhibitor, in Patients With Mild to Moderate Hypertension and Type 2 Diabetes Mellitus
Brief Title: A Comparison of Indapamide SR 1.5 mg With HCTZ 25 mg, in Combination With an ACE-inhibitor, in Patients With Mild to Moderate AHT and Type 2 DM
Acronym: AISHA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LaborMed Pharma S.A. (Industry)
Responsible Party: Professor Dragos Vinereanu, University and Emergency Hospital Bucharest, Cardiology Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RO-SCL-IQ v 1.0/04.07
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus
Keywords: blood tests; cardiac function; endothelial function; arterial function
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Hydrochlorothiazide; Indapamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide
- Indapamide SR (Experimental)
  Interventions: Drug: Indapamide

INTERVENTIONS:
Drug: Hydrochlorothiazide — orally, 25 mg, once a day, with Quinapril 10-40 mg, 6 months
  Other Names: Nefrix
  Arms: Hydrochlorothiazide
Drug: Indapamide — 1.5 mg SR, orally, once a day,with Quinapril 10-40 mg, 6 months
  Other Names: Indapamid LPH
  Arms: Indapamide SR

SUMMARY:
The aim of this study is to evaluate the effects of indapamide SR 1.5 mg on blood pressure, blood tests (glucose metabolism, lipids, minerals, and uric acid), cardiac function, endothelial and arterial function, by comparison with hydrochlorothiazide 25 mg, in patients with hypertension and type 2 diabetes mellitus. In order to achieve a better control of blood pressure in these patients, each diuretic treatments will be added to an ACE inhibitor (quinapril 10-40 mg/day). Therefore, eventually, the study will provide data on the comparison between combination indapamide SR 1.5 mg + quinapril versus hydrochlorothiazide 25 mg + quinapril.

DETAILED DESCRIPTION:
Hypertension treatment in patients with type 2 diabetes mellitus is still a difficult clinical problem. New European and American guidelines recommend a target blood pressure of less than 130/80 mmHg. Indeed, it was shown by the Hypertension Optimal Treatment study (HOT study) that reducing diastolic blood pressure to 81 mm Hg instead of 84 mm Hg, the number of major cardiovascular events is reduced by 51%. However, only 25% of the patients with hypertension and diabetes reach the target of 130/80 mm Hg in routine clinical practice. Therefore, combination therapy is always recommended (8, 9). This should include a diuretic; however, none of the two guidelines makes any recommendations regarding which is the best diuretic therapy in hypertensive patients with diabetes.

Indapamide is a diuretic with special characteristics, which was shown in experimental studies to provide cardio- and renal- protection in hypertensive patients. In the same time it has similar antihypertensive effects with amlodipine and hydrochlorothiazide. Intrinsic mechanisms are probably related to the antioxidant properties, and also to the action on the calcium channels. Moreover, when compared with hydrochlorothiazide, indapamide has no adverse effects on lipid metabolism and seems to have no negative impact on the renal function. However, a recent study in patients with hypertension and diabetes suggested no superiority of indapamide over hydrochorothiazide on different metabolic parameters. Therefore, new research looking in more detail to the comparison between the two diuretics is mandatory.

The aim of this study is to evaluate the effects of indapamide SR 1.5 mg on blood pressure, blood tests (glucose metabolism, lipids, minerals, and uric acid), cardiac function, endothelial and arterial function, by comparison with hydrochlorothiazide 25 mg, in patients with hypertension and type 2 diabetes mellitus. In order to achieve a better control of blood pressure in these patients, each diuretic treatments will be added to an ACE inhibitor (quinapril 10-40 mg/day). Therefore, eventually, the study will provide data on the comparison between combination indapamide SR 1.5 mg + quinapril versus hydrochlorothiazide 25 mg + quinapril.

The study will be conducted according to a Prospective, parallel, Randomized, active-controlled, Open, Blinded Endpoint evaluation (PROBE design), in one centre, in at least 50 male and female patients with mild to moderate hypertension and type 2 diabetes mellitus, for a total period of 18 months (12 months of enrollment and 6 months follow-up). Patients who meet the inclusion and exclusion criteria will be randomized 1:1 using a permuted block design. They will receive an ascending number from 1 to 50. The investigator(s) performing and analyzing the echocardiograms, and the central laboratory measuring the BNP blood tests will be blinded to the patient medication.

Patients will be randomized to either indapamide prolonged-release 1.5 mg/day or hydrochlorothiazide 25 mg/day, given orally. Quinapril will be added from the beginning of the study to allow consistent blood pressure control. Dose of quinapril will be titrated from 10 mg/day to 15 mg/day, and then to 20 mg/day, and up to 40 mg/day, as needed for the blood pressure control. The treatment will be administered to randomized patients for 6 months. Assignment of the study medication will be performed through randomization process. The patients will receive the medication from the Investigator/Co-investigator at every visit scheduled; they will be asked to return, at every visit scheduled, the unused medication and the empty boxes, in order to verify their compliance to the treatment. A treatment compliance of 80-120% is considered satisfactory for the study. If compliance is out of the limits mentioned above, the investigator can decide withdrawal of the patient from the study. In exceptional situations, the treatment can be interrupted for a period of maximum 3 days, without withdrawal of the patient from the study. The administration of the study medication will be documented in appropriate source documents and in the CRF and certified by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

Only diabetic patients presenting all of the following criteria should be enrolled into the study:

* Aged between 18 and 75 years .
* Daytime ambulatory blood pressure >135 and/or >85 mm Hg (only mild to moderate hypertension can be included in the study), and type 2 diabetes mellitus. The blood pressure monitoring device will be installed at visit 0 (Screening) and the conclusion of this monitoring will be evaluated at Visit1, before randomization.
* Sinus rhythm.
* Ability to understand the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the Investigator/Co-investigator, and to comply with the requirements of the study. Any anti-hypertensive medication will be stopped at least two weeks prior to randomisation.
* Informed written consent given before the initiation of the pre-study screening.

Exclusion Criteria:

* Secondary hypertension
* Severe hypertension ( ≥ 180 and/or ≥110 mm Hg); stage III hypertension (WHO classification)
* Symptoms of congestive heart failure (NYHA II - IV) or left ventricular global systolic dysfunction (EF < 40%)
* Ventricular aneurysm or extensive wall motion abnormalities
* Recent (< 6 months) myocardial infarction
* Recent (< 3 months) or planned coronary revascularization: PCI (percutaneous coronary intervention)/CABG (coronary artery by-pass graft)
* Severe valvular heart disease/congenital heart disease
* Hypertrophic cardiomyopathy
* Pericarditis
* Chronic cor pulmonale
* Recent (< 6 months) cerebrovascular ischemic symptoms (e.g. transient ischemic accident, prolonged reversible ischemic neurological deficit, stroke)
* Creatinine level >1.5 mg/dl for men or >1.4 mg/dl for women
* Pregnancy or patients who plan to become pregnant during the study period (only for female subjects).
* Breast-feeding woman
* Presence or history of relevant medical conditions, including: cancer, HIV, significant disease of the renal, hepatic, gastrointestinal, respiratory, endocrine, locomotor systems, or significant metabolic, haematological, neurological disorders
* History of hypersensitivity to indapamide, quinapril, thiazides or to any of the components of the products; contraindication to any of the study medications
* Significant acute illness within 14 days prior to randomisation
* Any history of drug or alcohol abuse, recent psychiatric disorder or use of psychotropic substances
* Any current condition or other disease known to interfere significantly with the absorption, distribution, metabolism or excretion of study drugs
* Current use of hormonal contraceptive drugs (only for female subjects); non-hormonal contraceptive measures have to be used, for female patients of childbearing potential, as follows: diaphragm, male condom, intrauterine device, tube ligation, selective tube occlusion procedure, or vasectomy of the partner
* Participation to another investigational study in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Better metabolic effects of indapamide SR 1.5 mg+quinapril by comparison with hydrochlorothiazide 25 mg+quinapril, in patients with hypertension and type 2 diabetes mellitus. | 6 months

SECONDARY OUTCOMES:
Better antihypertensive effects of indapamide SR 1.5 mg+quinapril by comparison with hydrochlorothiazide 25 mg+quinapril, in patients with hypertension and type 2 diabetes mellitus. | 6 months
Better effects on cardiac and arterial function of indapamide SR 1.5 mg+quinapril by comparison with hydrochlorothiazide 25 mg+quinapril, in patients with hypertension and type 2 diabetes mellitus | 6 months
Better safety of indapamide SR 1.5 mg+quinapril by comparison with hydrochlorothiazide 25 mg+quinapril, in patients with hypertension and type 2 diabetes mellitus | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Vinereanu, Professor, MD, PhD, Principal Investigator — Cardiology, University and Emergency Hospital, Bucharest, Romania
Locations (1):
- Cardiology, University and Emergency Hospital, Bucharest, Romania